CLINICAL TRIAL: NCT03235687
Title: A Prospective, Randomized Blinded, Shared Decision Impact Trial of the ExoDx Prostate (IntelliScore), EPI Test, in Men Presenting for Initial Biopsy.
Brief Title: Decision Impact Trial of the ExoDx Prostate (IntelliScore)
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Exosome Diagnostics, Inc. (Industry)
Collaborators: CareFirst BlueCross BlueShield (Unknown); Chesapeake Urology Research Associates (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Screening
Other Study IDs: ECT2017-002
Record Dates: First submitted 2017-07-28; First posted 2017-08-01 (Actual); Last update posted 2022-05-06 (Actual); Status verified 2022-05

CONDITIONS: Cancer of the Prostate
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Intervention Model Description: This is a prospective, randomized blinded, shared decision-impact and health-economic assessment study. 1000 appropriately screened consecutive patients seen during planning for a prostate biopsy will be enrolled. 500 patients will be randomized (blinded) to have the ExoDx Prostate (IntelliScore) test (Cohort A) and 500 (Cohort B) will proceed with conventional standard of care. At time of enrollment, neither the patient nor the urologist will be made aware of whether the patient will have an ExoDx Prostate (IntelliScore) test as part of their work-up. Cohort A EPI test results will be sent to the urologist for assessment and ultimately shared with the patient.
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Cohort A (Experimental): Patients randomized to Cohort A will receive ExoDx Prostate (IntelliScore) test results along with a post-ExoDx Prostate (IntelliScore) test result questionnaire to evaluate impact of test results in the biopsy decision process, utility, ease of understanding and work-flow implementation.
  Interventions: Diagnostic Test: ExoDx Prostate (IntelliScore)
- Cohort B (No Intervention): Patients randomized to Cohort B will proceed with conventional standard of care.

INTERVENTIONS:
Diagnostic Test: ExoDx Prostate (IntelliScore) — ExoDx Prostate (IntelliScore) is a non-invasive, urinary 3-gene expression validated test in which the results of the assay are adjunctive to the ordering physician's clinical judgment and work-up of the patient in the determination of whether a prostate needle biopsy is necessary. The ExoDx Prostate (IntelliScore) was clinically validated to discriminate patients with higher grade prostate cancer from those with more indolent lower grade cancer and benign disease.
  Other Names: EPI
  Arms: Cohort A

SUMMARY:
The purpose of this research study is to investigate the utility of a validated urine test which predicts the likelihood of high grade prostate cancer on an initial prostate biopsy.

DETAILED DESCRIPTION:
Primary Objective(s)

1. Evaluate performance of the ExoDx Prostate(IntelliScore) (EPI) to reduce the number of initial prostate biopsies by greater than or equal to 15% for men with an elevated Prostate-Specific Antigen 2-10ng/mL presenting for a biopsy in consultation with their urologist.
2. Compare performance of both the ExoDx Prostate(IntelliScore) 15.6 and 20 cut-points with respect to the biopsy decision process.
3. Assess physician satisfaction with the ExoDx Prostate(IntelliScore) report including test result presentation, graphics and interpretation.
4. Assess urologist / patient satisfaction for ease of understanding test results and role on biopsy decision process.

Secondary Objectives

1. Determine the medical economic impact of the ExoDx Prostate(IntelliScore) test in the prostate biopsy decision process.
2. Correlation of the ExoDx Prostate(IntelliScore) score with the actual biopsy result by utilizing the Receiver Operating Characteristic of the Area Under Curve for discriminating high-grade (greater than or equal to Gleason Score 7, International Society of Urological Pathology 2 and 3) from low-grade (Gleason Score 6, International Society of Urological Pathology 1) and benign disease on initial prostate needle biopsy.

ELIGIBILITY:
Inclusion Criteria:

* 50 years of age
* Clinical suspicion for prostate cancer
* Elevated Prostate-specific antigen between: 2.0 - 10 ng/ mL
* No clinical history of a prior negative biopsy

Exclusion Criteria:

* History of prior prostate biopsy.
* Use of medications or hormones that are known to affect serum Prostate-specific antigen levels within 3-6 months of study enrollment.
* Clinical symptoms of urinary tract infection (including prostatitis) at the time of enrollment.
* History of prostate cancer.
* History of invasive treatments for benign prostatic hypertrophy (Benign Prostatic Hyperplasia) or lower urinary track symptoms within 6 months of study enrollment.
* Known hepatitis (all types) and/or HIV documented in patient's medical record.
* Patients with history of concurrent renal/bladder tumors.

Min Age: 50 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Must be male to screen for prostate cancer
Enrollment: 1000 (Estimated)
Dates: Start 2017-07-19 (Actual); Primary Completion 2018-09-01 (Actual); Study Completion 2023-09-29 (Estimated)

PRIMARY OUTCOMES:
Evaluate performance of the ExoDx Prostate(IntelliScore) | 6 Months
  Evaluate performance of the ExoDx Prostate(IntelliScore) to reduce the number of initial prostate biopsies by greater than or equal to 15% for men with an elevated prostate specific antigen between 2-10ng/mL presenting for a biopsy in consultation with their urologist.

CONTACTS AND LOCATIONS:
Overall Officials: Roger Tun, Study Director — Exosome Diagnostics, Inc.; Ronald F Tutrone, MD, Principal Investigator — Chesapeake Urology Research Associates
Locations (1):
- Chesapeake Urology Research Associates, Towson, Maryland, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Tutrone R, Donovan MJ, Torkler P, Tadigotla V, McLain T, Noerholm M, Skog J, McKiernan J. Clinical utility of the exosome based ExoDx Prostate(IntelliScore) EPI test in men presenting for initial Biopsy with a PSA 2-10 ng/mL. Prostate Cancer Prostatic Dis. 2020 Dec;23(4):607-614. doi: 10.1038/s41391-020-0237-z. Epub 2020 May 7. PMID 32382078
- [Derived] Tutrone R, Lowentritt B, Neuman B, Donovan MJ, Hallmark E, Cole TJ, Yao Y, Biesecker C, Kumar S, Verma V, Sant GR, Alter J, Skog J. ExoDx prostate test as a predictor of outcomes of high-grade prostate cancer - an interim analysis. Prostate Cancer Prostatic Dis. 2023 Sep;26(3):596-601. doi: 10.1038/s41391-023-00675-1. Epub 2023 May 16. PMID 37193776
- [Derived] Kretschmer A, Tutrone R, Alter J, Berg E, Fischer C, Kumar S, Torkler P, Tadigotla V, Donovan M, Sant G, Skog J, Noerholm M. Pre-diagnosis urine exosomal RNA (ExoDx EPI score) is associated with post-prostatectomy pathology outcome. World J Urol. 2022 Apr;40(4):983-989. doi: 10.1007/s00345-022-03937-0. Epub 2022 Jan 27. PMID 35084544